CLINICAL TRIAL: NCT04004091
Title: Prenatal Administration of Oral Spermine Promotes Maturation of Premature Fetal Gut Epithelial Tight Junction: Experimental Study on Oryctolagus Cuniculus
Brief Title: Prenatal Administration of Spermine Promotes Maturation of Premature Fetal Gut Epithelial Tight Junction: Experimental Study on Fetal Rabbit
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: dr. Riana Pauline Tamba, SpB(K)BA (Other)
Responsible Party: Sponsor-Investigator, dr. Riana Pauline Tamba, SpB(K)BA, Consultant Pediatric Surgeon, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: tight junction, spermine
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Premature Birth; NEC
Keywords: Premature Birth; Spermine; Necrotizing Enterocolitis; Tight Junction
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Spermine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- 24-Day Spermine Group (Experimental): Subjects are given prenatal spermine (20 mg per body weight) during 24 days of pregnancy. On day 24 pregnancy is terminated and intestinal tissue sample is taken to be examined.
  Interventions: Biological: Spermine
- 26-Day Spermine Group (Experimental): Subjects are given prenatal spermine (20 mg per body weight) during 26 days of pregnancy. On day 26 pregnancy is terminated and intestinal tissue sample is taken to be examined.
  Interventions: Biological: Spermine
- 28-Day Spermine Group (Experimental): Subjects are given prenatal spermine (20 mg per body weight) during 28 days of pregnancy. On day 28 pregnancy is terminated and intestinal tissue sample is taken to be examined.
  Interventions: Biological: Spermine
- 24-Day Non Spermine Group (No Intervention): Subjects are not given any intervention. On day 24 pregnancy is terminated and intestinal tissue sample is taken to be examined.
- 26-Day Non Spermine Group (No Intervention): Subjects are not given any intervention. On day 26 pregnancy is terminated and intestinal tissue sample is taken to be examined.
- 28-Day Non Spermine Group (No Intervention): Subjects are not given any intervention. On day 28 pregnancy is terminated and intestinal tissue sample is taken to be examined.

INTERVENTIONS:
Biological: Spermine — Spermine is a polyamine. It is an organic molecule that is involved in cellular metabolism and development.
  Arms: 24-Day Spermine Group; 26-Day Spermine Group; 28-Day Spermine Group

SUMMARY:
Infections, particularly on the gastrointestinal tract, has been known to be one of the leading causes of death in preterm infants. This is due to the immaturity of the intestinal epithelial cells. Recent studies have shown that polyamines have a role on the development of cells during embryonal phase. By this experimental study, the investigators would like to evaluate the administration of spermine on the maturation of premature fetal gut epithelial tight junction.

DETAILED DESCRIPTION:
This experimental study is conducted with minimum 24 subjects which divided into 6 groups; 1) 24-days pregnant and is given prenatal spermine, 2) 26-days pregnant and is given prenatal spermine, 3) 28-days pregnant and is given prenatal spermine, 4) 24-days pregnant and is not given prenatal spermine, 5) 26-days pregnant and is not given prenatal spermine, and 6) 28-days pregnant and is not given prenatal spermine. At the end of desired pregnancy period, hysterectomy is done and fetus are born. From each parent subject, three fetal samples are chosen using a random sampling. Intestinal tissues are taken from each fetal sample to be examined. Several data will be collected i.e. occludin, β-catenin, and β-actin, as well as histological morphologies.

ELIGIBILITY:
Inclusion Criteria:

* Intestinal tissue of fetal rabbit that is prematurely alive

Exclusion Criteria:

* Intestinal tissue of fetal rabbit that is dead before termination
* Intestinal tissue of fetal rabbit, in which the parent died before termination

Ages: 24 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occludin | 2 weeks
  Measurement of occludin (ng/mg protein) from intestinal tissue sample is assessed using Rabbit Occludin ELISA Kit
β-catenin | 2 weeks
  Measurement of β-catenin (pg/mg protein) from intestinal tissue sample is assessed using Rabbit β-Catenin ELISA Kit
β-actin | 2 weeks
  Measurement of β-actin (ng/mg protein) from intestinal tissue sample is assessed using β-Actin ELISA Kit

SECONDARY OUTCOMES:
Histologic Findings | 2 weeks
  Identifying the development of epithelial tight junction cells based on the morphologic findings of the villi structure, including Goblet cells' distribution, enterocytes, enteroendocrine cells, and crypts.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo National Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Wettere WH, Willson NL, Pain SJ, Forder RE. Effect of oral polyamine supplementation pre-weaning on piglet growth and intestinal characteristics. Animal. 2016 Oct;10(10):1655-9. doi: 10.1017/S1751731116000446. Epub 2016 Mar 21. PMID 26997172
- [Background] Peulen O, Gharbi M, Powroznik B, Dandrifosse G. Differential effect of dietary spermine on alkaline phosphatase activity in jejunum and ileum of unweaned rats. Biochimie. 2004 Jul;86(7):487-93. doi: 10.1016/j.biochi.2004.06.002. PMID 15308338
- [Background] Peulen O, Dandrifosse G. Spermine-induced maturation in wistar rat intestine: a cytokine-dependent mechanism. J Pediatr Gastroenterol Nutr. 2004 May;38(5):524-32. doi: 10.1097/00005176-200405000-00012. PMID 15097442
- [Background] Greco S, Niepceron E, Hugueny I, George P, Louisot P, Biol MC. Dietary spermidine and spermine participate in the maturation of galactosyltransferase activity and glycoprotein galactosylation in rat small intestine. J Nutr. 2001 Jul;131(7):1890-7. doi: 10.1093/jn/131.7.1890. PMID 11435503
- [Background] Peulen O, Pirlet C, Klimek M, Goffinet G, Dandrifosse G. Comparison between the natural postnatal maturation and the spermine-induced maturation of the rat intestine. Arch Physiol Biochem. 1998 Feb;106(1):46-55. doi: 10.1076/apab.106.1.46.4392. PMID 9783060
- [Background] Wery I, Deloyer P, Dandrifosse G. Effects of a single dose of orally-administered spermine on the intestinal development of unweaned rats. Arch Physiol Biochem. 1996;104(2):163-72. doi: 10.1076/apab.104.2.163.12886. PMID 8818200
- [Background] Harada E, Hashimoto Y, Syuto B. Orally administered spermine induces precocious intestinal maturation of macromolecular transport and disaccharidase development in suckling rats. Comp Biochem Physiol A Physiol. 1994 Nov;109(3):667-73. doi: 10.1016/0300-9629(94)90208-9. PMID 8529008